CLINICAL TRIAL: NCT03010774
Title: Identifying At-Risk Patients and Predicting Deterioration of In-Patients Using Continuous Heart Rate, Respiratory Rate, and Movement Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: EarlySense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB13-0885
Record Dates: First submitted 2016-12-14; First posted 2017-01-05 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Risk Stratification (Experimental): Study participants will be risk stratified according to the eCART scoring algorithm each night. If they are stratified as low risk, they will not receive routine nighttime spot-check vital signs unless indicated by a change in patient status or monitor alarm.
  Interventions: Behavioral: Risk Stratification
- Control - Usual Care (Active Comparator): Study participants will be woken at night for routine nighttime spot-check vital signs regardless of patient disease severity or risk.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Risk Stratification — Every night, subjects will be risk stratified into low-risk or medium- to high-risk using a physiologic risk score, eCART. Subjects who meet the low-risk criteria will not be woken up for routine nighttime vitals (typically at midnight and at 4 am). However, subjects will continue to be woken up for laboratory draws, procedures, or treatments as per usual. Subjects who are medium- to high-risk will continue to be woken up at night for routine nighttime vitals. Alarms for all subjects, including low-risk subjects, will continue to alert nurses in real-time. If the primary nurse of a low-risk subject is alerted of an alarm, the nurse will have to go into the subject's room to turn off the alarm and therefore check on the patient.
  Arms: Intervention - Risk Stratification
Behavioral: Usual Care — The subject will continue to receive routine vital sign measurements and charting, standard for the ward or according to the physician orders, including routine spot-check vital signs, regardless of risk level.
  Arms: Control - Usual Care

SUMMARY:
Currently, all patients in the hospital are woken up throughout the night to check for vital signs, no matter how sick they are. The investigators are doing this study to determine whether skipping routine vital sign checks at night improves participant sleep quality and satisfaction without increasing the risk of adverse events.

DETAILED DESCRIPTION:
The purpose of this study is:

1. To determine the correlation between subjective and objective sleep quality measures.
2. To compare the objective and subjective measures of sleep quality and satisfaction between the intervention group and the control group.
3. To compare the adverse event rates in the intervention group and the control group, defined as ICU transfer or cardiac arrest occurring within 24 hours of risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Hospitalized on study unit

Exclusion Criteria:

* Inability to provide consent
* Non-English speaking
* Order for physical wound checks
* Order for cardiac telemetry monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | 5 days
  Pittsburgh Sleep Quality Index
Sleep Quality | 5 days
  Karolinska Sleep Log
Sleep Quality | 5 days
  Potential Hospital Sleep Disruptions and Noises Questionnaire

SECONDARY OUTCOMES:
Adverse Event Rate | within 24 hours of risk stratification
  ICU transfer or cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Dana P Edelson, MD, MS, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States